CLINICAL TRIAL: NCT03959176
Title: The Effect of Brimonidine on Intraocular Pressure When Dilating Routine Patients, Pressure Control and Pupil Effects
Brief Title: The Effect of Brimonidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00058366
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2020-07

CONDITIONS: Intraocular Pressure
Keywords: Brimonidine; Pupil Effects
MeSH Terms: interventions — Brimonidine Tartrate; Tropicamide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): The right eye will receive a sham drop followed by 1 drop of Tropicamide 1%/Phenylephrine 2.5% five minutes after the sham drop is administered. A one minute wait will occur followed by a second drop of Tropicamide 1%/Phenylephrine 2.5%.
  The left eye will receive 2 drops of Brimonidine 0.2% followed by a five minute wait time. One drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a one minute wait time. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered.
  Interventions: Drug: Brimonidine; Drug: Tropicamide; Drug: Phenylephrine Ophthalmic Product
- Group 2 (Experimental): The right eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered followed by a 15 second wait after which a sham drop will be administered.
  The left eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a 15 second wait after which 2 drops of Brimonidine will be administered.
  Interventions: Drug: Brimonidine; Drug: Tropicamide; Drug: Phenylephrine Ophthalmic Product

INTERVENTIONS:
Drug: Brimonidine — 2 drops administered once in the left eye in both study arms
  Other Names: Alphagan; Mirvaso
Drug: Tropicamide — 1 drop administered at two different times points in both eyes in both study arms
  Other Names: Mydriacyl
Drug: Phenylephrine Ophthalmic Product — 1 drop administered at two different time points in both eyes in both study arms

SUMMARY:
This study will evaluate whether pre-treating patients with Brimonidine 0.2% before and/or after dilating the pupils will help to control the changes in intraocular pressure often seen when using dilating drops. The study will also evaluate the effects of different sequences of administering dilating drops along with Brimonidine on pupil size and reactivity.

DETAILED DESCRIPTION:
Intraocular pressure (IOP) can fluctuate due to various external factors such as exercise, medications, and eye movements. Although it is considered natural for IOP to fluctuate daily, prolonged increases in IOP can be harmful. Sustained elevated IOP has been linked to optic nerve damage and glaucoma. Mydriatic drops routinely given to dilate pupils in patients in need of an eye exam have been known to increase IOP. In practice, a combination of drugs are used to achieve pupil dilation needed for routine eye exams or in perioperative situations. The use of Tropicamide 1% and Phenylephrine 2.5% are known to be safe and effective options for dilating the pupils when used in conjunction with one another, but these drugs can increase IOP. Drugs such as Brimonidine, a selective alpha-2 agonist, are known to reduce IOP through several different methods. This study seeks to understand the effects of Brimonidine used along with Tropicamide and Phenylephrine to control IOP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Females of childbearing potential must agree to use a reliable method of birth control while participating in the study.

Exclusion Criteria:

* Diabetic
* Have a history of glaucoma
* Have a history of iris trauma
* Have a history of eye surgery except for LASIK or PRK
* Pregnant
* Anisocoria (unequal pupils)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Walter, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Overall results will be shared, but individual participant data will not be available.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Group 1: The right eye will receive a sham drop followed by 1 drop of Tropicamide 1%/Phenylephrine 2.5% five minutes after the sham drop is administered. A one minute wait will occur followed by a second drop of Tropicamide 1%/Phenylephrine 2.5%.
  The left eye will receive 2 drops of Brimonidine 0.2% followed by a five minute wait time. One drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a one minute wait time. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered.
  Brimonidine: 2 drops administered once in the left eye in both study arms
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
- Group 2: The right eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered followed by a 15 second wait after which a sham drop will be administered.
  The left eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a 15 second wait after which 2 drops of Brimonidine will be administered.
  Brimonidine: 2 drops administered once in the left eye in both study arms
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
Period: First Eye Exam
Arm/Group | Group 1 | Group 2
Started | 7; 7 Eyes (Right eyes) | 6; 6 Eyes (Right eyes)
Completed | 7; 7 Eyes (Right eyes) | 6; 6 Eyes (Right eyes)
Not Completed | 0; 0 Eyes | 0; 0 Eyes
Period: Opposite Eye Exam
Arm/Group | Group 1 | Group 2
Started | 7; 7 Eyes (Left eyes) | 6; 6 Eyes (Left eyes)
Completed | 7; 7 Eyes (Left eyes) | 6; 6 Eyes (Left eyes)
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (.7) | 23.7 (1.5) | 23.25 (.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: To observe how differing the sequence of administration of Tropicamide 1%/Phenylephrine 2.5% and Brimonidine 0.2% influences intraocular pressure.
Time Frame: Baseline (Pre drop administration)
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Units Other Than Participants: Eyes
Groups:
- Group 1 Right Eye: The right eye will receive a sham drop followed by 1 drop of Tropicamide 1%/Phenylephrine 2.5% five minutes after the sham drop is administered. A one minute wait will occur followed by a second drop of Tropicamide 1%/Phenylephrine 2.5%.
  Tropicamide: 1 drop administered at two different times points in both left and right eyes
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both left and right eyes
- Group 1 Left Eye: The left eye will receive 2 drops of Brimonidine 0.2% followed by a five minute wait time. One drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a one minute wait time. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered.
  Brimonidine: 2 drops administered once in the left eye
  Tropicamide: 1 drop administered at two different times points in both left and right eyes
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both left and right eyes
- Group 2 Right Eye: The right eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered followed by a 15 second wait after which a sham drop will be administered.
  Tropicamide: 1 drop administered at two different times points in both the left and right eyes.
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both the left and right eyes.
- Group 2 Left Eye: The left eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a 15 second wait after which 2 drops of Brimonidine will be administered.
  Brimonidine: 2 drops administered once in the left eye
  Tropicamide: 1 drop administered at two different times points in both the left and right eyes.
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points both the left and right eyes.
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
millimeters of mercury (mmHg) | 15.4 (2.4) | 16.3 (2.4) | 16.5 (1.5) | 16.7 (1.3)

2. Primary Outcome: Intraocular Pressure
Description: as for outcome 1
Time Frame: 15 minutes post drop administration
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mmHg | 15.3 (2.0) | 13.1 (1.5) | 13.5 (1.7) | 15.0 (1.2)

3. Primary Outcome: Intraocular Pressure
Description: as for outcome 1
Time Frame: 30 minutes post drop administration
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Group 2 Right Eye: The right eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered followed by a 15 second wait after which a sham drop will be administered.
  Tropicamide: 1 drop administered at two different times points in both the left and right eyes.
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both the left and right eyes.
  The left eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a 15 second wait after which 2 drops of Brimonidine will be administered.
  Brimonidine: 2 drops administered once in the left eye in both study arms
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
mmHg | 14.6 (1.7) | 12.3 (1.5) | 14.3 (1.8) | 14.8 (1.4)

4. Primary Outcome: Intraocular Pressure
Description: as for outcome 1
Time Frame: 1 hour post drop administration
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mmHg | 15.1 (2.0) | 12.4 (1.8) | 13.5 (2.0) | 13.2 (1.9)

5. Primary Outcome: Intraocular Pressure
Description: as for outcome 1
Time Frame: 2 hour post drop administration
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mmHg | 14.3 (1.7) | 11.9 (1.4) | 12.7 (1.0) | 14.2 (1.3)

6. Primary Outcome: Intraocular Pressure
Description: as for outcome 1
Time Frame: 4 hour post drop administration
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mmHg | 12.4 (1.7) | 9.3 (1.3) | 11.0 (1.2) | 13.7 (1.8)

7. Secondary Outcome: Pupil Size
Description: Pupil size measurement
Time Frame: Baseline (Pre drop administration)
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
millimeter (mm) | 3.7 (.4) | 3.7 (.4) | 4.1 (.4) | 4.1 (.4)

8. Secondary Outcome: Pupil Size
Description: Pupil size measurement.
Time Frame: 15 minutes post drop administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mm | 7.9 (.4) | 8.6 (.3) | 7.6 (.4) | 7.9 (.3)

9. Secondary Outcome: Pupil Size
Description: Pupil size measurement
Time Frame: 30 minutes post drop administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mm | 8.3 (.4) | 9.6 (.2) | 8.1 (.4) | 8.8 (.4)

10. Secondary Outcome: Pupil Size
Description: Pupil size measurement.
Time Frame: 1 hour post drop administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mm | 8.9 (.3) | 8.9 (.3) | 8.3 (.4) | 9.1 (.2)

11. Secondary Outcome: Pupil Size
Description: Pupil size measurement.
Time Frame: 2 hours post drop administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mm | 8.7 (.3) | 8.7 (.3) | 7.8 (.5) | 8.6 (.3)

12. Secondary Outcome: Pupil Size
Description: Pupil size measurement
Time Frame: 4 hours post drop administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (Eyes) | 7 | 7 | 6 | 6
mm | 7.6 (.4) | 7.6 (.4) | 6.7 (.5) | 7.6 (.7)

13. Secondary Outcome: Pupil Reaction to Light
Description: Pupil reaction to light will be measured as none (0), poor (1) or brisk (2).
Time Frame: Baseline (Pre drop administration)
Population: Data only collected for Right Eye in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 6
score on a scale | 2 (0) | 2 (0)

14. Secondary Outcome: Pupil Reaction to Light
Description: Pupil reaction to light will be measured as none (0), poor (1) or brisk (2).
Time Frame: 15 minutes post drop administration
Population: Data only collected for Right Eye in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 6
score on a scale | 0 (0) | 0 (0)

15. Secondary Outcome: Pupil Reaction to Light
Description: Pupil reaction to light will be measured as none (0), poor (1) or brisk (2).
Time Frame: 30 minutes post drop administration
Population: Data only collected for Right Eye in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 6
score on a scale | 0 (0) | 0 (0)

16. Secondary Outcome: Pupil Reaction to Light
Description: Pupil reaction to light will be measured as none (0), poor (1) or brisk (2).
Time Frame: 1 hour post drop administration
Population: Data only collected for Right Eye in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 6
score on a scale | 0 (0) | 0 (0)

17. Secondary Outcome: Pupil Reaction to Light
Description: Pupil reaction to light will be measured as none (0), poor (1) or brisk (2).
Time Frame: 2 hours post drop administration
Population: Data only collected for Right Eye in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 6
score on a scale | 0 (0) | 0 (0)

18. Secondary Outcome: Pupil Reaction to Light
Description: Pupil reaction to light will be measured as none (0), poor (1) or brisk (2).
Time Frame: 4 hours post drop administration
Population: Data only collected for Right Eye in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 6
score on a scale | 1 (0) | 1 (0)

ADVERSE EVENTS:
Time Frame: baseline through hour 4
Groups:
- Group 1 Right Eye: The right eye will receive a sham drop followed by 1 drop of Tropicamide 1%/Phenylephrine 2.5% five minutes after the sham drop is administered. A one minute wait will occur followed by a second drop of Tropicamide 1%/Phenylephrine 2.5%.
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
- Group 1 Left Eye: The left eye will receive 2 drops of Brimonidine 0.2% followed by a five minute wait time. One drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a one minute wait time. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered.
  Brimonidine: 2 drops administered once in the left eye in both study arms
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
- Group 2 Right Eye: The right eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will be administered followed by a 15 second wait after which a sham drop will be administered.
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
- Group 2 Left Eye: The left eye will receive 1 drop of Tropicamide 1%/Phenylephrine 2.5% followed by a one minute wait. A second drop of Tropicamide 1%/Phenylephrine 2.5% will then be administered followed by a 15 second wait after which 2 drops of Brimonidine will be administered.
  Brimonidine: 2 drops administered once in the left eye in both study arms
  Tropicamide: 1 drop administered at two different times points in both eyes in both study arms
  Phenylephrine Ophthalmic Product: 1 drop administered at two different time points in both eyes in both study arms
- All Group 1 Participants; All Group 2 Participants: The whole participant including all body systems.
Arm/Group | Group 1 Right Eye | Group 1 Left Eye | Group 2 Right Eye | Group 2 Left Eye | All Group 1 Participants | All Group 2 Participants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03959176/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT03959176/ICF_000.pdf